CLINICAL TRIAL: NCT06768671
Title: An Open-label, Single-arm Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous Sonelokimab in Adolescents Aged ≥12 to ≤17 Years at the Time of Study Inclusion With Active Moderate to Severe Hidradenitis Suppurativa
Brief Title: An Open-label, Single-arm Study to Evaluate Pharmacokinetics and Safety of Subcutaneous Sonelokimab in Adolescents With Moderate to Severe Hidradenitis Suppurativa (VELA-TEEN)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M1095-HS-304
Record Dates: First submitted 2024-11-29; First posted 2025-01-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration; Anti-Inflammatory Agents; Sonelokimab; Nanobody; Apocrine Gland Disease
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Sweat Gland Diseases; Skin Diseases; Skin Diseases, Bacterial; Suppuration | interventions — sonelokimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sonelokimab (Experimental): Subjects will receive sonelokimab 120mg subcutaneously (SC) as an induction regimen of 4 doses, followed by sonelokimab SC every 4 weeks maintenance dose starting at Week 8
  Interventions: Drug: Sonelokimab

INTERVENTIONS:
Drug: Sonelokimab — Open label

SUMMARY:
This is a study to evaluate the pharmacokinetic (PK) and safety of sonelokimab in adolescent patients with HS.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between ≥12 and ≤17 years of age at the time of signing the informed consent.
2. Participants who are diagnosed with HS as determined by the investigator and have a history of signs and symptoms of HS for ≥6 months before signing the informed consent.
3. Participants who have moderate to severe HS as determined by the refined Hurley staging (Stages IB and IC, IIB and IIC, and III).
4. Participants who have had an inadequate response to appropriate systemic antibiotics for treatment of HS .
5. Participants must be up to date with age-appropriate vaccine requirements 8 weeks prior to entry in the study.
6. Participants with a body weight of ≥ 40 kg.

Exclusion Criteria:

1. Participants with a known hypersensitivity to sonelokimab or any of its excipients.
2. Participants with a draining fistula count of ≥20 at the Screening Visit.
3. Participants with any other active skin disease or condition that may, in the opinion of the investigator, interfere with the assessment of HS.
4. Participants with underlying conditions that, in the opinion of the investigator, potentially compromise the participant and/or places the participant at unacceptable risk.
5. Participants who have history or concurrent clinically significant medical conditions or any other reason, including any physical, psychological, or psychiatric condition, that in the opinion of the investigator would compromise the safety or interfere with participation in the study, would make the participant an unsuitable candidate to receive study drug, or would put the participant at risk.
6. Participants with any other skin disease or other medical condition that in the opinion of the investigator would interfere with an accurate assessment of clinical symptoms of HS.
7. Participants with a confirmed or suspected diagnosis of inflammatory bowel disease.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of sonelokimab in adolescents | Week 24
  PK (trough concentrations) of sonelokimab over 24 weeks of treatment
Adverse events (AEs) following treatment with sonelokimab in adolescents | Week 24
  Incidence, relatedness, severity and seriousness of all AEs over 24 weeks of treatment from baseline
Discontinuation of sonelokimab treatment due to AEs | Week 24
  Number of participants discontinued from sonelokimab treatment due to AE over 24 weeks of treatment from baseline
Clinically significant changes in clinical laboratory parameters | Week 24
  Number of participants with clinically significant changes in hematology, biochemistry and urinalysis from baseline
Clinically significant changes in vital signs | Week 24
  Number of participants with clinically significant changes in vital signs from baseline
Clinically significant changes in standard 12-lead electrocardiogram (ECG) intervals | Week 24
  Number of participants with clinically significant changes in 12-lead ECG intervals from baseline

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR)75 | Week 24
  Percentage of participants achieving a HiSCR75 response over time
Hidradenitis Suppurativa Clinical Response (HiSCR) 50 | Week 24
  Percentage of participants achieving a HiSCR50 response over time
International Hidradenitis Suppurativa Severity Score System (IHS4) | Week 24
  Absolute change in IHS4 score over time
Children's Dermatology Life Quality Index (CDLQI) | Week 24
  Percentage of participants achieving a CDLQI total reduction of ≥2.5 over time among participants with a baseline CDLQI ≥2.5
Numerical Rating Scale (NRS) 30 | Week 24
  Percentage of participants achieving a ≥30% reduction and a ≥2-unit reduction over time in the NRS30 for pain in PGA among participants with a baseline NRS ≥3

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Clinical Site, North Little Rock, Arkansas
  - Clinical Site, Stanford, California
  - Clinical Site, Washington D.C., District of Columbia
  - Clinical Site, Hollywood, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Macon, Georgia
  - Clinical Site, Sandy Springs, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Columbus, Indiana
  - Clinical Site, Murray, Kentucky
  - Clinical Site, Waterford, Michigan
  - Clinical Site, Fargo, North Dakota
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Dallas, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Norfolk, Virginia
  - Clinical Site, Seattle, Washington